CLINICAL TRIAL: NCT02532777
Title: The Research of Standard Diagnosis and Treatment for Henoch-Schonlein Purpura Nephritis in Children
Brief Title: The Research of Standard Diagnosis and Treatment for HSPN in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Aihua Zhang, Hospital vice president, Nanjing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZhang
Record Dates: First submitted 2015-08-20; First posted 2015-08-26 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Henoch-Schoenlein Purpura Nephritis
MeSH Terms: interventions — Prednisone; Mycophenolic Acid; Leflunomide; Angiotensin-Converting Enzyme Inhibitors; benazepril; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prednisone & Cyclophosphamide (Experimental): Drug: prednisone & cyclophosphamide & Angiotensin-converting enzyme inhibitor(ACEI).
  Prednisone: 2mg/kg/d (the maximum dose is 60mg) for 6-8 weeks, then two-thirds of the two day's dose qod.
  cyclophosphamide: 0.1mg/kg. Angiotensin-converting enzyme inhibitor(ACEI): 0.2-0.3mg/kg/d. Methylprednisolone: the children with above 50% crescent in renal biopsy.
  Interventions: Drug: Prednisone; Drug: Cyclophosphamide(CTX); Drug: Angiotensin-converting enzyme inhibitor(ACEI); Drug: Methylprednisolone
- Prednisone & Mycophenolate mofetil (Experimental): Drug: prednisone & mycophenolate mofetil & Angiotensin-converting enzyme inhibitor(ACEI).
  Prednisone: 2mg/kg/d (the maximum dose is 60mg) for 6-8 weeks, then two-thirds of the two day's dose qod.
  mycophenolate mofetil: 25mg/kg/d bid (the maximum dose is 1.5g/d). Angiotensin-converting enzyme inhibitor(ACEI): 0.2-0.3mg/kg/d. Methylprednisolone: the children with above 50% crescent in renal biopsy.
  Interventions: Drug: Prednisone; Drug: Mycophenolate mofetil(MMF); Drug: Angiotensin-converting enzyme inhibitor(ACEI); Drug: Methylprednisolone
- Prednisone & Leflunomide (Experimental): Drug: prednisone & leflunomide & Angiotensin-converting enzyme inhibitor(ACEI). Prednisone: 2mg/kg/d (the maximum dose is 60mg) for 6-8 weeks, then two-thirds of the two day's dose qod.
  Leflunomide: give patients the induction dose 1mg/kg/d for three days (the total dose is under 40mg/kg)，then give the maintaining dose 0.5mg/kg/d.
  Angiotensin-converting enzyme inhibitor(ACEI): 0.2-0.3mg/kg/d. Methylprednisolone: the children with above 50% crescent in renal biopsy.
  Interventions: Drug: Prednisone; Drug: Leflunomide(LEF); Drug: Angiotensin-converting enzyme inhibitor(ACEI); Drug: Methylprednisolone

INTERVENTIONS:
Drug: Prednisone
Drug: Cyclophosphamide(CTX)
  Arms: Prednisone & Cyclophosphamide
Drug: Mycophenolate mofetil(MMF)
  Arms: Prednisone & Mycophenolate mofetil
Drug: Leflunomide(LEF)
  Arms: Prednisone & Leflunomide
Drug: Angiotensin-converting enzyme inhibitor(ACEI)
  Other Names: Lotensin
Drug: Methylprednisolone

SUMMARY:
This study is performed to evaluate the efficacy and safety of various measures in the treatment of HSPN in children.

DETAILED DESCRIPTION:
Henoch-Schonlein purpura nephritis (HSPN) is one of the most common complications of Henoch-Schonlein purpura, and has become one of the main causes of chronic kidney disease in children. However, the diagnosis and treatment of HSPN is still based on the clinical experience, lacking of evidence-based support. This study is performed to explore the biological marker for early prediction of the prognosis and evaluate the efficacy and safety of various measures in the treatment of HSPN in children.

The patients who are proved to get HSPN by renal biopsy will be given prednisone 2mg/kg/d, and randomized to receive cyclophosphamide pulse i.v.,mycophenolate mofetil p.o. or leflunomide p.o., we will follow up them for about 2.5 years and compare the efficacy and safety of these measures by monitoring several indexes.

ELIGIBILITY:
Inclusion Criteria:

* Renal biopsy proved HSPN Proteinuria ≥ 50 mg/kg/d

Exclusion Criteria:

* The children with congenital diseases Proteinuria < 50 mg/kg/d

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Disappearance of proteinuria | 30 mo
  The proteinuria is < 150mg/d

SECONDARY OUTCOMES:
Disappearance of hematuria | 30 mo
  The number of red blood cells is < 3 in each high power field of vision
Renal function | 30 mo
  The glomerular filtration rate is normal

CONTACTS AND LOCATIONS:
Overall Officials: Aihua Zhang, M.D., Study Chair — Department of Nephrology, Nanjing children's hospital
Locations (1):
- Nanjing Children's Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hahn D, Hodson EM, Craig JC. Interventions for preventing and treating kidney disease in IgA vasculitis. Cochrane Database Syst Rev. 2023 Feb 28;2(2):CD005128. doi: 10.1002/14651858.CD005128.pub4. PMID 36853224